CLINICAL TRIAL: NCT02922296
Title: Glucose Metabolism in Sickle Cell Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Victor Gordeuk, Director Sickle Cell Center, University of Illinois at Chicago
Other Study IDs: 2015-0366
Record Dates: First submitted 2016-07-31; First posted 2016-10-04 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Diabetes Mellitus
MeSH Terms: conditions — Anemia, Sickle Cell; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be stored temporarily in the laboratory of the Principal Investigator at the University of Illinois at Chicago, long term storage of specimens will be at the UIC Biobank. The research data will be stored in a locked file cabinet in the PI's research office. The patient's name or other identifying data will not be revealed, except to those directly involved in this study.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to better understand how the body handles sugars glucose and fats, such as cholesterol and triglycerides in sickle cell disease, and what puts certain persons at risk to develop diabetes. This understanding may help us to find new treatments to control blood sugar and prevent diabetes in people with and without sickle cell disease (SCD).

In this research, DNA and RNA will be isolated from blood cells. DNA will be used to find genes that cause or protect from diabetes, high cholesterol and high triglyceride, and RNA will be used for studies designed to find out how genes are doing their job of eventually producing proteins.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is due to homozygosity for a Glu6Val mutation in HBB (sickle cell anemia; hemoglobin SS) or to compound heterozygous forms like hemoglobin SC disease and hemoglobin S-β thalassemia. Past studies suggested a low prevalence of diabetes in patients with SCD.10 Improvements in treatment and care have increased the life span of patients. This, along with the wide availability of high calorie diets and increasing adiposity in SCD raises that possibility that the prevalence of diabetes is increasing in SCD. Our study is designed to characterize the changes in metabolism that occur in sickle cell disease and to identify clinical, genetic and genomic risk factors for the development of diabetes. Our hypothesis is that non-overweight subjects with SCD have relative protection from diabetes and metabolic syndrome, but that those individuals who do become overweight have a dramatic increase in the rates of diabetes and metabolic syndrome. Lean SCD subjects will not have simply a neutral, but an overtly anti-diabetic phenotype (e.g. better glucose tolerance and lower metabolic syndrome markers). The two main study aims are as follows; Aim 1. Define the metabolic status of adult SCD subjects according to normal or increased BMI.

Aim 2. Determine genetic and genomic predictors of overweight, metabolic syndrome and diabetes in SCD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Major sickling genotype (hemoglobin SS, Sbeta0-thalassemia, SOarab, SDpunjab)
* Age >35 years
* BMI <25 kg/m2 or >26 kg/m2
* Steady state, defined as >two weeks from a hospitalization for vaso-occlusive crisis, infection or surgery and not requiring immediate parenteral medication for pain control
* Fasting state (>8 hours since ingesting food or medication for diabetes)

Exclusion Criteria:

* Patients receiving insulin therapy
* Acute inflammatory or infectious illness or injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult sickle cell disease subjects, with or without diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-05-01; Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic status of adult SCD subjects | through study completion, approximately one year after subject participation
  The investigator will use the ATP III guidelines for definition of metabolic syndrome. A combination of any three of the following criteria will lead to the designation of metabolic syndrome:
  * waist circumference >102 cm (men) or >88 cm (women)
  * triglycerides ≥150 mg/dL
  * HDL cholesterol <40 mg/dL (men) or <50 mg/dL (women)
  * blood pressure ≥130/≥85 mg/dL (or recorded diagnosis of hypertension and use of antihypertensives)
  * fasting glucose ≥110 mg/dL (or diagnosis of diabetes and use of anti-diabetic medications)

SECONDARY OUTCOMES:
Genetic and genomic predictors in SCD subjects | through study completion, approximately one year after subject participation
  This will be accomplished by DNA linkage analysis and/or mutation analysis. In addition RNA will be isolated from from PBMCs and fractions of platelets, granulocytes and reticulocytes. The investigators will analyze the expression of transcripts to determine if alterations can explain the clinical observations.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Gordeuk, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No